CLINICAL TRIAL: NCT02736305
Title: An Open-Label, Single-Arm Phase 2 Clinical Trial Of Regorafenib in Patients With Multiply Recurrent Epithelial Ovarian Cancer
Brief Title: Use of Regorafenib in Recurrent Epithelial Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC OV-01
Record Dates: First submitted 2015-10-13; First posted 2016-04-13 (Estimated); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Ovarian Neoplasms
Keywords: ovarian; regorafenib; platinum resistant; clear cell; endometrioid
MeSH Terms: conditions — Ovarian Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Regorafenib (Experimental): Patients will receive Regorafenib 120mg once daily, with consideration for dose escalation to 160mg if there are no toxicities
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — Once a day for 21 days in a 28 days cycle
  Other Names: Stivarga

SUMMARY:
Regorafenib is an oral multikinase inhibitor that blocks the activity of kinases involved in angiogenesis (VEGFR 1,2,3 and TEK), oncogenesis (KIT, Ret Proto-Oncogene (RET), Raf-1 Proto-Oncogene, Serine/Threonine Kinase (RAF1) and BRAF) and tumour growth (PDGFR and FGFR). Epithelial ovarian cancer (EOC) cell lines frequently express high levels of vascular endothelial growth factor (VEGF) and in vivo preclinical studies evaluating Regorafenib have shown promising activity in ovarian cancer. In the clinic, anti-angiogenesis therapy with bevacizumab (a monoclonal antibody to VEGF) has already emerged as an important cornerstone in the management of ovarian cancer both as part of frontline adjuvant treatment and as second-line therapy for platinum-sensitive recurrent disease. Whilst Regorafenib has been FDA approved for the treatment of patients with metastatic colorectal cancer who have failed prior bevacizumab, it's role in the management of ovarian cancer remains to be defined.

DETAILED DESCRIPTION:
STUDY OBJECTIVES

The objective of this study is to evaluate the efficacy and safety of regorafenib at a dose of 120mg daily for 21 days out of every 28 day cycle in Asian females with multiply recurrent EOC.

Primary Endpoint:

Investigator assessed progression free survival (PFS)

Secondary Endpoints:

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent obtained before any study specific procedures. Subjects must be able to understand and willing to sign a written informed consent.
2. Patients with histologically and/or cytologically confirmed epithelial ovarian carcinoma (serous, clear cell, endometrioid, mucinous, mixed, carcinosarcoma and others), fallopian tube and primary peritoneal carcinoma.
3. Progressive disease following 2 or more prior cytotoxic chemotherapy. Patients may have received prior treatment with bevacizumab.
4. Age ≥ 21 years old
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
6. Life expectancy greater than 3 months
7. Measurable disease by RECIST 1.1 OR non measurable but evaluable disease such as ascites and pleural effusions attributable to disease or radiologic abnormalities that did not meet RECIST criteria AND a pre-treatment serum Ca-125 level greater than or equal to 2 times the upper limit of normal on 2 occasions at least 1 week apart OR pre treatment Ca-125 level greater or equal to 2 times the upper limit of normal on 2 occasions at least 1 week apart and non evaluable, non measurable disease.
8. Adequate bone marrow function as shown by: absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelet count ≥ 100 x 109/L and haemoglobin (Hb) > 9 g/dl. Blood transfusion to meet the inclusion criteria will not be allowed.
9. Adequate liver function as assess by: total bilirubin ≤ 1.5 x upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x ULN or ≤ 5.0 x ULN if liver metastases are present.
10. Adequate renal function as assessed by serum creatinine ≤ 1.5 x ULN and glomerular filtration rate (GFR) ≥ 30 ml/min according to Cockcroft-Gault formula.
11. Systolic blood pressure ≤ 160 mmHg.
12. Women of childbearing potential and men must agree to use adequate contraception since signing of the informed consent form until at least 3 months after the last study drug administration. The investigator or a designated associate is requested to advise the subject on how to achieve adequate birth control. Adequate contraception is defined in the study as any medically recommended method (or combination of methods) as per standard of care.
13. International normalized ratio (INR) ≤ 1.5 x ULN and partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless receiving treatment with therapeutic anticoagulation. Patients being treated with anticoagulant e.g. heparin will be allowed to participate provided no prior evidence of an underlying abnormality in these parameters exists.

Exclusion Criteria:

1. Patients who are receiving any other investigational agents.
2. Previous assignment to treatment during this study. Subjects permanently withdrawn from study treatment participation will not be allowed to re-enter the study.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition used in the study.
4. Prior treatment with regorafenib.
5. Previous or concurrent cancer that is distinct in primary site of histology from EOC within the last 5 years EXCEPT for curatively treated cervical cancer in situ, non melanoma skin cancer and superficial bladder tumours [Ta (non invasive tumour), Tis (carcinoma in situ) and T1 (tumour invades lamina propria)].
6. Patients with known brain metastases.
7. Uncontrolled inter-current illness including, but not limited to, on going or active infection (> Grade 2 NCI CTCAE v 4.00), symptomatic congestive heart failure (≥ New York Heart Association (NYHA) class 2), unstable angina pectoris, new onset angina (begun within the last 3 months), myocardial infarction less than 6 months before, cardiac arrhythmia requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted), pre existing poorly controlled hypertension (systolic blood pressure > 160mmHg or diastolic pressure > 90 mmHg despite optimal medical management), history of abdominal fistula, history of gastrointestinal perforation and signs or symptoms of bowel obstruction.
8. Subjects with phaeochromocytoma.
9. Other concurrent severe and/or uncontrolled concomitant medical conditions that could cause unacceptable safety risk or compromise compliance with the protocol.
10. Patients unable to swallow orally administered medication and patients with impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of either study drug (e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhoea, malabsorption syndrome).
11. Patients who have undergone major surgery, open biopsy of significant traumatic injury ≤ 28 days prior to starting study drug.
12. Patient with bowel resection within the past 1 year.
13. Patients with a past history of bowel perforation and abdominal fistula; patients with a recent history of bowel resection (within the past 12 months) and/or patients with symptoms of radiological evidence of active bowel obstruction.
14. Extended field radiotherapy within 4 weeks or limited field radiotherapy within 2 weeks prior to randomization. Patients must have recovered from all therapy related toxicities. The site of previous radiotherapy should have evidence of progressive disease if this is the only site of disease.
15. Patients with venous thromboembolism disease or pulmonary embolism within 6 months before start of study medication (except for adequately treated catheter-related venous thrombosis occurring more than one month before the start of study medication).
16. Arterial thrombotic event including transient ischaemic attack (TIA), cerebrovascular accident (CVA) and peripheral arterial embolus within the last 6 months before start of study medication.
17. Subjects with evidence or history of any bleeding diathesis irrespective of severity.
18. Non-healing wound, ulcer or bone fracture.
19. Known history of human immunodeficiency virus (HIV) infection.
20. Subjects with seizure disorder requiring medication.
21. History of organ allograft.
22. Renal failure requiring haemo- or peritoneal dialysis.
23. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
24. Interstitial lung disease with on-going signs and symptoms at the time of informed consent.
25. Systemic anticancer therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy and hormonal therapy during this trial or within 4 weeks (or 6 weeks for nitrosurea, antibodies or mitomycin-C) prior to starting study drug or who have not recovered from side effects of such therapy.
26. Pregnant or breast-feeding in females. Women of childbearing potential must have a pregnancy test performed a maximum of 7 days before start of treatment, and a negative result must be documented before start of treatment.
27. Inability to attend or comply with treatment of follow-up scheduling.
28. Persistent proteinuria > 3.5g/24 hours measured by urine protein-creatinine ratio from a random urine sample
29. Any haemorrhage or bleeding event ≥ CTCAE Grade 3 within 4 weeks prior to the start of study medication
30. Active hepatitis B or C, or chronic hepatitis B or C requiring treatment with antiviral therapy

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
Investigator assessed progression free survival (PFS) | 30 days after the last dose of regorafenib

SECONDARY OUTCOMES:
Overall survival (OS) | 30 days after the last dose of regorafenib
Overall tumour response rate (ORR) as per Gynecological Cancer Intergroup (GCIG) and RECIST v1.1 criteria | 30 days after the last dose of regorafenib
Treatment Emergent Adverse Events | 30 days after the last dose of regorafenib
  During the study period, patients will undergo evaluations for safety and drug tolerability.
  * Unexpected and expected toxicities including Hand Foot Syndrome, Liver dysfunction, Hypertension, Bleeding, Nausea and Diarrhoea
  * Death

OTHER OUTCOMES:
Health Related Quality of Life (HRQoL) | 30 days after the last dose of regorafenib
Maximum Plasma Concentration [Cmax] | 30 days after the last dose of regorafenib
Area Under the Curve (AUC) | 30 days after the last dose of regorafenib

CONTACTS AND LOCATIONS:
Overall Officials: Wen Yee Chay, MBBS, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided